CLINICAL TRIAL: NCT02222350
Title: A Phase 2, Placebo-controlled, Double-blind Study of DS-8500a in Patients With Type 2 Diabetes
Brief Title: Phase 2 Study of DS-8500a in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DS8500-A-J201
Record Dates: First submitted 2014-08-18; First posted 2014-08-21 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2015-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — firuglipel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- DS-8500a 10mg once daily (Experimental): 10mg DS-8500a tablet given orally once daily
  Interventions: Drug: 10mg DS-8500a tablet
- DS8500a 75 mg once daily (Experimental): 75mg DS-8500a tablet given orally once daily
  Interventions: Drug: 75mg DS-8500a tablet
- placebo to match DS-8500a tablet (Placebo Comparator): placebo matching DS-8500a tablet
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: 10mg DS-8500a tablet
  Arms: DS-8500a 10mg once daily
Drug: 75mg DS-8500a tablet
  Arms: DS8500a 75 mg once daily
Drug: placebo
  Arms: placebo to match DS-8500a tablet

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of DS-8500a compared with placebo in Japanese patients with Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the efficacy and safety of DS-8500a 10 mg and 75 mg administered orally, once daily, for 28 days, compared with placebo, in Japanese patients with Type 2 Diabetes Mellitus in a double-blind, placebo-controlled parallel-group design. The primary endpoint is the change in 24-hour weighted mean glucose at day 28 from baseline. The safety, pharmacokinetics, and pharmacodynamics of DS-8500a will be evaluated as well.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 20 years at the time of informed consent
* Japanese patients with type 2 diabetes
* Patients who have HbA1c ≥ 7.0% and < 10.0% if untreated with antidiabetic agent.
* Patients who have HbA1c ≥ 6.5% and < 9.5% if treated with antidiabetic agent.

Exclusion Criteria:

* Patients aged ≥ 70 years at the time of informed consent
* Patients with a history of type 1 diabetes or diabetic ketoacidosis
* Patients receiving or requiring treatment with insulin
* Patients with a body mass index (BMI) of < 18.5 kg/m2 or ≥ 35.0 kg/m2
* Patients with an estimated glomerular filtration rate (eGFR), < 45 mL/min per 1.73 m2
* Patients with fasting plasma glucose ≥ 240 mg/dL

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-07; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
change in 24-hour weighted mean blood glucose | Day -1 (baseline) to Day 28

SECONDARY OUTCOMES:
change in 24 hour weighted mean blood glucose | Day -1 (baseline) to Day 14
change in blood fasting plasma glucose level | Day -1 (baseline) to Days 7, 14, 21, 28
change in blood plasma glucose level | Day -1 (baseline) to Days 14 and 28
  Change in the parameter at Day 14 or 28 from Day -1
change in blood insulin level | Day -1 (baseline) to Days 14 and 28
  Change in the parameter at Day 14 or 28 from Day -1
change in blood C-peptide level | Day -1 (baseline) to Days 14 and 28
  Change in the parameter at Day 14 or 28 from Day -1
change in blood active GLP-1 level | Day -1 (baseline) to Days 14 and 28
  Change in the parameter at Day 14 or 28 from Day -1
change in blood PYY level | Day -1 (baseline) to Days 14 and 28
  Change in the parameter at Day 14 or 28 from Day -1
change in blood HbA1c level | Day -1 (baseline) to Days 14 and 28
  Change in the parameter at Day 14 or 28 from Day -1
change in blood glycoalbumin level | Day -1 (baseline) to Days 14 and 28
  Change in the parameter at Day 14 or 28 from Day -1
Number of subjects experiencing adverse events as a measure of safety | Day -1 (baseline) to Day 28
  Number of subjects experiencing adverse events
pharmacokinetic profile of DS-8500a | Day -1 (baseline) to Day 28
  Pharmacokinetic profile of DS-8500a in Japanese subjects with type 2 diabetes mellitus. i.e. Tmax, Cmax, AUC, t1/2
change in postprandial plasma glucose level | Day -1 (baseline) to Days 14 and 28
  Change in postprandial plasma glucose level (2 hours after a meal) at Day 14 or 28 from Day -1

CONTACTS AND LOCATIONS:
Locations (1):
- Heishinkai Medical Group Incorporated OCROM Clinic, Kasuga, Osaka, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Inagaki N, Chou HS, Tsukiyama S, Washio T, Shiosakai K, Nakatsuka Y, Taguchi T. Glucose-lowering effects and safety of DS-8500a, a G protein-coupled receptor 119 agonist, in Japanese patients with type 2 diabetes: results of a randomized, double-blind, placebo-controlled, parallel-group, multicenter, phase II study. BMJ Open Diabetes Res Care. 2017 Sep 29;5(1):e000424. doi: 10.1136/bmjdrc-2017-000424. eCollection 2017. PMID 29071087